CLINICAL TRIAL: NCT03534973
Title: Prevention of Experimental Ultraviolet Induced Apoptosis in Explanted Human Lens Epithelial Cells Enriched With Caffeine: a Pilot Study
Brief Title: Prevention of UV- Induced Apoptosis by Caffeine
Acronym: Caff2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Caff2
Record Dates: First submitted 2018-04-30; First posted 2018-05-23 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Cataract
Keywords: Cataract; Caffeine
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine intake (Active Comparator): Caffeine is given orally prior to cataract surgery
  Interventions: Other: Caffeine intake
- No caffeine intake (Sham Comparator): Caffeine is not given orally prior to cataract surgery
  Interventions: Other: No caffeine intake

INTERVENTIONS:
Other: Caffeine intake — Cataract surgery in eyes with prior caffeine intake
  Arms: Caffeine intake
Other: No caffeine intake — Cataract surgery in eyes without prior caffeine intake
  Arms: No caffeine intake

SUMMARY:
Investigate if caffeine accumulation in human lens epithelial cells after oral caffeine intake is sufficient to prevent from experimental ultraviolet radiation induced apoptosis

DETAILED DESCRIPTION:
Caffeine is a worldwide consumed dietary constituent. It occurs in a variety of beverages such as coffee, tea, soft drinks and cocoa beverages, and in chocolate-based food products. In the United States there is a reported average intake of caffeine of 200 mg/d in 80 % of adults corresponding to the amount in two 5-ounce cups of coffee or four sodas. A new interest for caffeine in ophthalmology emerged with the observation that caffeine inhibits cataractogenesis.

Cataract is the leading cause of blindness worldwide and until now there is no approved drug to prevent cataract. UVR-B radiation has been identified as one of the major risk factors for age related cataract. In vitro, Varma showed that caffeine preserves ATP levels and GSH levels in the lens when exposed to UVR-B and further maintains the state of transparency in the lens. Varma moreover hypothesized that its protective effect in the lens is due to its ability to scavenge reactive oxygen species (ROS) and to suppress elevation of toxic microRNAs and consequent gene silencing. In the galactosemic rat model, Varma demonstrated that topical caffeine in vivo inhibited the formation of galactose cataract and prevented apoptosis of lens epithelial cells.

A further study presented evidence that topical caffeine also prevents in vivo UVR-B induced cataract and inhibits apoptosis of lens epithelial cells. The investigators estimated the protection factor (PF) of caffeine to 1.23. The PF is identical to PF for sunscreens; the ratio between the threshold dose of the toxic agent and the threshold dose without the toxic agent. The PF observed for topically applied caffeine was higher than the PF observed for perorally administered vitamin E (PF: 1.14) and vitamin C (PF: 1) , respectively. Only the Grx gene provides a higher PF (PF 1.3). This strongly supports that caffeine has an important antioxidant capacity in vivo.

Up to 99 % of caffeine is gastrointestinally absorbed and pharmacokinetics are comparable after oral and i.v. administration. In the liver, caffeine is metabolized by hepatic enzymes belonging to the cytochrome P-450 family, mainly CYP1A2. Major metabolites like 1-methylxanthine and 1-methyl uric acid were reported to still have significant antioxidant activity. Recently, a study confirmed the protective effect of coffee combined with additional antioxidant dietary against age-related cataract. Its hydrophobic properties allow caffeine passage over all biological membranes. A further study found that caffeine after oral intake accumulates in the lens epithelium.

The lens epithelium plays a major role in balancing water, ions and the metabolic homeostasis. Additionally, the germinative cells in the lens epithelium generate a reservoir for lens fiber cell generation. UVR-B radiation is absorbed by proteins and DNA in the lens epithelium and underlying lens fibres, causing damage to the cells. When epithelial cells are damaged, lens growth and transparency is disturbed. Michael et al. demonstrated the appearance of apoptotic lens cells after in vivo exposure to UVR-B with transmission electron microscopy. No necrotic cells were found at threshold dose. We found a peak of Apoptosis hours after UVR-B exposure.

The present study aims to investigate if caffeine accumulation in human lens epithelial cells after oral caffeine intake is sufficient to prevent from experimental ultraviolet radiation induced apoptosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Cataract
* Patients who chose pseudoanalgesia technique for cataract surgery before recruitment process
* Written informed consent prior to surgery

Exclusion Criteria:

* Age < 21 years
* Beverages containing caffeine (such as Coffee, Coca Cola, energy drinks, black or green tea) and dark chocolate consumption 1 week before surgery
* Pseudoexfoliation syndrome of the lens
* Systolic hypertension of >160 at the day of surgery
* Pregnancy (pregnancy test will be taken in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of apoptotic and viable lens epithelial cells from eyes with and without oral caffeine intake | 12 months
  Using a cell apoptosis and viability assay the number of apoptotic and viable lens epithelial cells is counted under a fluorescence microscope

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided